CLINICAL TRIAL: NCT06829095
Title: Personalized Nutrition Counseling to Improve the Nutritional Status of Esophageal Cancer or Head and Neck Cancer Patients Undergoing Concurrent Chemoradiotherapy
Brief Title: Personalized Nutrition Counseling and Nutritional Status of Esophageal Cancer and HNSCC Patients Undergoing CCRT
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsuan-Chih Kuo, Professor Attending Physicians, Chang Gung Memorial Hospital
Other Study IDs: 202300755B0
Record Dates: First submitted 2023-11-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer; Personalized Nutrition
Keywords: Personalized nutrition; Esophageal cancer; Concurrent chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: Under the same condition of nutritional supplements in both the experimental group and the control group,the investigators explore the changes in the quality of life and nutritional status of the subjects by evaluating with the nutrition Index (PG-SGA) and quality of life (EORTC QLQ-C30 questionnaire Taiwan version) questionnaire evaluation and recode the basic physical data, including body weight, grip strength, body muscle fat composition.
- experimental: Dietitians consult with participants which invited to be the experimental group and follow up weekly through communication software (Line) or telephone remote methods. Dietitians provide the dietary advice base on the guidance of the cancer diet principles, and give on assessment and diet adjustments.Under the same condition of nutritional supplements in both the experimental group and the control group,the investigators explore the changes in the quality of life and nutritional status of the subjects by evaluating with the nutrition Index (PG-SGA) and quality of life (EORTC QLQ-C30 questionnaire Taiwan version) questionnaire evaluation and recode the basic physical data, including body weight, grip strength, body muscle fat composition.

SUMMARY:
The purpose of the study is to improve the nutritional status of esophageal cancer patients undergoing concurrent chemoradiotherapy by the personalized nutrition counseling.Dietitians consult with participants which invited to be the experimental group and follow up weekly through communication software (Line) or telephone remote methods. Dietitians provide the dietary advice base on the guidance of the cancer diet principles, and give on assessment and diet adjustments. At the same time, Under the same condition of nutritional supplements in both the experimental group and the control group, the investigators explore the changes in the quality of life and nutritional status of the subjects by evaluating with the nutrition Index (PG-SGA) and quality of life (EORTC QLQ-C30 questionnaire Taiwan version) questionnaire evaluation and recode the basic physical data, including body weight, grip strength, body muscle fat composition. Therefore, investigators conducted this study to appoint dietitian to arrange personalized nutrition consultation for esophageal cancer patients to improve the nutritional status of these patients.

DETAILED DESCRIPTION:
Approximately 60-85% of esophageal cancer patients present with malnutrition at diagnosis (1). Malnutrition, defined as body weight loss of more than 10% over the previous 6 months is associated with treatment response and survival (2). Around 38% of esophageal cancer patients are managed with curative intent in the form of neoadjuvant chemotherapy or chemoradiotherapy followed by esophagectomy (3). Individuals are at increased risk of malnutrition arising from disease related symptoms and neoadjuvant treatment. Nutritional status serves as an important risk factor for major complications after operation (4) Therefore, assessment of nutritional status should be undertaken for all esophageal cancer patients, especially for those who are planned to receive esophagectomy (5). The nutritional assessment includes hand grip for muscle mass (6), body composition for lean body mass and sarcopenia (7), body mass index- body weight loss grade (BMI-BWL grade) for generalized nutrition status (8). These tools are needed to be integrated and individualized to esophageal cancer patients to improve outcome. Therefore, investigators conducted this trial to appoint dietitian to arrange personalized nutrition consultation for esophageal cancer patients to improve the nutritional status of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically and CT confirmed esophageal cancer or head and neck cancer
2. CCRT therapy
3. ECOG performance status grade≦2
4. agree to participate the trial
5. over 18 years
6. no pregnant

Exclusion Criteria:

1. have two or more cancers
2. gastrointestinal tract cannot function
3. NYHA class 4
4. abnormal liver and kidney function
5. Abnormal bone marrow hematopoiesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal cancer or head and neck cancer patients undergoing concurrent chemoradiotherapy
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
BMI in kg/m^2-W1 | baseline
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
BMI in kg/m^2-W2 | 2nd week
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
BMI in kg/m^2-W3 | 3rd week
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
BMI in kg/m^2-W4 | 4th week
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
BMI in kg/m^2-W5 | 5th week
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
BMI in kg/m^2-W6 | 6th week
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
BMI in kg/m^2-W12 | 12th week
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
BMI in kg/m^2-W18 | 18th week
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
BMI in kg/m^2-W30 | 30th week
  Document of participant's BMI and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W1 | baseline
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W2 | 2nd week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W3 | 3rd week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W4 | 4th week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W5 | 5th week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W6 | 6th week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W12 | 12th week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W18 | 18th week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
hand grip in kg-W30 | 30th week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W1 | baseline
  Document of participant's body fat and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W2 | 2nd week
  Document of participant's hand grip and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W3 | 3rd week
  Document of participant's body fat and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W4 | 4th week
  Document of participant's body fat and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W5 | 5th week
  Document of participant's body fat and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W6 | 6th week
  Document of participant's body fat and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W12 | 12th week
  Document of participant's body fat and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W18 | 18th week
  Document of participant's body fat and evaluating the effectiveness of nutritionist health education nutritional status
body fat in kg-W30 | 30th week
  Document of participant's body fat and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W1 | baseline
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W2 | 2nd week
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W3 | 3rd week
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W4 | 4th week
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W5 | 5th week
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W6 | 6th week
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W12 | 12th week
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W18 | 18th week
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
muscle weight in kg-W30 | 30th week
  Document of participant's muscle weight and evaluating the effectiveness of nutritionist health education nutritional status
CTC cell number counting in number-W1 | baseline
  Document of participant's CTC cell number counting and evaluating the effectiveness of nutritionist health education nutritional status
CTC cell number counting in number-W6 | 6th week
  Document of participant's CTC cell number counting and evaluating the effectiveness of nutritionist health education nutritional status
CTC cell number counting in number-W18 | 18th week
  Document of participant's CTC cell number counting and evaluating the effectiveness of nutritionist health education nutritional status

SECONDARY OUTCOMES:
Abridged Patient-Generated Subjective Global Assessment, aPG-SGA Questionnaire W1 | baseline
  nutrition consultation and do the SGA questionnaire(the minimum value is 1 and the maximum value is 36. The higher scores mean a worse outcome) for recoding and improving the nutritional status of participants.
Abridged Patient-Generated Subjective Global Assessment, aPG-SGA Questionnaire W3 | 3th week
  nutrition consultation and do the SGA questionnaire(the minimum value is 1 and the maximum value is 36. The higher scores mean a worse outcome) for recoding and improving the nutritional status of participants.
Abridged Patient-Generated Subjective Global Assessment, aPG-SGA Questionnaire W6 | 6th week
  nutrition consultation and do the SGA questionnaire(the minimum value is 1 and the maximum value is 36. The higher scores mean a worse outcome) for recoding and improving the nutritional status of participants.
aPG SGA Questionnaire W18 | 18th week
  nutrition consultation and do the SGA questionnaire(the minimum value is 1 and the maximum value is 36. The higher scores mean a worse outcome) for recoding and improving the nutritional status of participants.
SGA-Questionnaire W30 | 30th week
  nutrition consultation and do the SGA questionnaire(the minimum value is 1 and the maximum value is 36. The higher scores mean a worse outcome) for recoding and improving the nutritional status of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Chih Kuo, Study Director — Division of Oncology, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, New Taipei City, Taiwan